CLINICAL TRIAL: NCT02552537
Title: Integrated Approaches to Food Allergen and Allergy Risk Management: iFAAM: The Impact of Proton-pump Inhibitors (Antacids) on Threshold Dose Distributions
Brief Title: iFAAM: The Impact of Proton-pump Inhibitors (Antacids) on Threshold Dose Distributions
Acronym: iFAAM-PPI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University of Nebraska Lincoln (Other); Region Hovedstadens Apotek (Other Government); University of Manchester (Other); Hospital San Carlos, Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KEK 2015-0380
Record Dates: First submitted 2015-09-14; First posted 2015-09-17 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Omeprazole; Mannitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omeprazole (Active Comparator): patients will take Omeprazole 40mg, in capsules, once a day, during five days before walnut challenge
  Interventions: Drug: Omeprazole
- Placebo (Sham Comparator): patients will take Mannitol, in capsules, once a day, during five days before walnut challenge
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omeprazole — patients with walnut allergy will be exposed during 5 days before food challenge with Omeprazole
  Other Names: Omeprazol Sandoz eco Kps 40
  Arms: Omeprazole
Drug: Placebo — patients with walnut allergy will be exposed during 5 days before food challenge with Placebo
  Other Names: Mannitol
  Arms: Placebo

SUMMARY:
In patients with a walnut allergy double blind placebo controlled food challenge with walnut will be combined with the intake of proton pump inhibitor (PPI) or with placebo to assess the impact of PPI on threshold level and on clinical manifestation.

DETAILED DESCRIPTION:
1. detailed case history, blood sampling and prick testing with different foods will performed.
2. double blind food provocation with with three meals containing either placebo or walnut in walnut allergic patients will be performed.
3. the provocation will be combined with the intake of drug (omeprazole) or placebo (mannitol) blinded in capsules.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent, history of walnut allergy,minimum age 18 years

Exclusion Criteria:

* • Known hypersensitivity or allergy to Omeprazole, other proton pump inhibitors, mannitol, ingredients of placebo meal

  * Drugs not allowed during the study due to proved interaction with Omeprazole: Digoxin, Clopidogrel, Methotrexate, Antiretroviral drugs, Diazepam, Cilostazol, Phenytoin, Warfarin (R-Warfarin) and other Vitamin K antagonists, Phenytoin, Tacrolimus, Clarithromycin, voriconazole, Rifampicin and Hypericum
  * Drugs not allowed due to interference with the food challenge (or shortest interval between last treatment and food challenge)
* corticosteroids systemically (2 weeks)
* antihistamines (3 days) except hydroxyzine (10 days)
* ketotifen (2 weeks)
* betablocker (1 day)
* angiotensin converting enzyme (ACE) inhibitors (2 days)
* omalizumab (2 months)

  * Women who are pregnant or breast feeding
  * Intention to become pregnant during the course of the study
  * Lack of safe contraception, defined as: female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices
  * Please note that female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
  * Uncontrolled asthma, forced expiratory volume <70% predicted value
  * Acute allergic disease
  * Chronic urticaria
  * Mastocytosis
  * Other clinically significant concomitant disease states (major organic or infectious diseases, e.g., renal failure, hepatic dysfunction, cardiovascular disease, acute febrile infection),
  * Known or suspected non-compliance, drug or alcohol abuse,
  * Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
  * Participation in another study with investigational drug within the 30 days preceding and during the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
amount of walnuts that induces an allergic reaction assessed in milligram | up to 18 months
  The amount of walnut which induces an allergic reaction in walnut allergic patients will be assessed in milligram by titrated challenges under concommitant intake of therapeutic doses of omeprazole versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Clare Mills, Prof, PhD, Study Chair — University Manchester
Locations (2):
- Hospital Clinico San Carlos, Madrid, Spain
- University Hospital Zurich, Zurich, Switzerland